CLINICAL TRIAL: NCT07210502
Title: Comparing the Side Effects of Low Dose Rate Brachytherapy Against Ultra-Hypofractionated Radiotherapy Using Spacer Gel Treatment in Men With Cambridge Prognostic Groups (CPG) 1 to 3 (NCCN Low to Intermediate Risk) Prostate Cancer
Brief Title: Side Effects of Low Dose Rate Brachytherapy and Ultra-hypofractionated Radiotherapy in Low to Intermediate Risk Prostate Cancer
Acronym: LDR BURST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LDR BURST Trial
Record Dates: First submitted 2025-06-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Prostate Adenocarcinoma
Keywords: low dose rate brachytherapy; Stereotactic Body Radiation Therapy; rectal spacer gel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 4D low dose rate brachytherapy (Active Comparator): Insertion of iodine -125 radioactive seeds in the prostate gland. Prescription dose 145 Gy. Permanent placement of seeds under general anaesthesia and real time image guidance. Post brachytherapy insertion of Barrigel (rectal space gel).
  Interventions: Radiation: 4D Low Dose Rate Prostate Brachytherapy
- Ultra-hypofractionated Radiotherapy (Active Comparator): Stereotactic Body Radiation Therapy (SBRT).Prescription dose 36.25 Gy given in 5 fractions over 1-2 weeks (i.e. daily or alternate daily) delivered on linear accelerator. All patients will have fiducial markers inserted prior to their treatment together with insertion of Barrigel (rectal space gel).
  Interventions: Radiation: Ultra-hypofractionated Radiotherapy

INTERVENTIONS:
Radiation: 4D Low Dose Rate Prostate Brachytherapy — Permanent implantation of radioactive seeds in the prostate gland which slowly deposit half their dose approximately every 60 days. Prescription dose 145 Gy.
  Arms: 4D low dose rate brachytherapy
Radiation: Ultra-hypofractionated Radiotherapy — The prescription dose is 36.25 Gy given in 5 fractions over 1-2 weeks (i.e. daily or alternate daily at department discretion) delivered on linear accelerator
  Arms: Ultra-hypofractionated Radiotherapy

SUMMARY:
The LDR BURST trial will compare the side effects of two radiotherapy treatments for men with localised prostate cancer. The first treatment is 4D low dose rate brachytherapy where small radioactive seeds are inserted into the prostate gland under ultrasound guidance. A computerised tomography scan is subsequently performed to check seed positioning. Patients usually return home the same day. The seeds emit their radiation over several months before losing their activity.

Stereotactic radiotherapy, an alternative treatment, is a form of external radiation using precise high energy x-rays to target the prostate gland. It is delivered in 5 treatment sessions on alternate days; the full treatment course is completed within 2 weeks.

Stereotactic radiotherapy has recently been approved by the National Health Service following successful results in international trials demonstrating it is safe and effective to give external radiotherapy in five treatment sessions. Delivering a higher dose in each treatment fraction is known as 'ultra-hypofractionation'. Before the treatment, men will undergo a minor procedure, typically under local anaesthetic, to have metallic markers inserted into the prostate to improve visibility of the prostate gland when planning and delivering the treatment.

The side effects of both the radiation treatments are similar. Common side effects include bladder issues, such as needing to urinate more often and having a slower urine flow. Patients might also experience more frequent and looser bowel movements, occasionally with a little blood. Symptoms usually improve over time. Additionally, some men might have trouble achieving or maintaining an erection after radiation treatment, this can often be managed with medications.

Both of the treatments use ionising radiation to destroy the prostate cancer cells which may cause cancer many years or decades after exposure. The chances of this happening are the same whether taking part in this trial or not.

A protective gel, called Barrigel, will be inserted into the space between the prostate gland and the rectum increasing the distance between them. This significantly reduces the dose of radiation to the rectum. The gel can be inserted at the same time as the brachytherapy seed or fiducial marker insertion. The gel is slowly reabsorbed following treatment over the next 3 to 6 months.

The trial will randomly assign 110 men to each radiation treatment to compare their side effects. There is a 50% chance the patient will be assigned to brachytherapy and 50% chance of stereotactic radiotherapy. Patients will be asked to complete four questionnaires prior to starting treatment and at regular time points following treatment. They will be telephoned every 4 weeks for the first 2 months to check on side effects, followed by a face-to-face appointment at 3 months, and a PSA blood test, and then followed up at regular intervals for 5 years.

DETAILED DESCRIPTION:
The hypothesis of the study is that treatment-related toxicity after Stereotactic Body Radiotherapy (SBRT) is not significantly different to that after Low Dose Rate (LDR) Brachytherapy. SBRT is an economically attractive strategy that is not invasive but requires multiple hospital visits (one visit per fraction, currently a minimum of 5 visits) whereas LDR Brachytherapy only requires one treatment visit. Both treatment options have independently shown excellent control of prostate cancer with low toxicity but high-quality evidence from a randomised controlled study with sufficient follow up on toxicity and efficiency comparing the two treatments is lacking.

Patients suitable for the trial will be highlighted at their local prostate cancer multidisciplinary team (MDT) at Royal Surrey County Hospital, Frimley Park Hospital, East Surrey Hospital & Ashford and St Peters Hospital (All hospitals are members of the Royal Surrey National Health Service (NHS)Trust). Patients deemed eligible for all radical treatment options for their prostate cancer (surgery or radiotherapy), will be reviewed by the surgical and oncology team as per standard of care management. Should the patient express an interest in radiation treatment and be willing to be randomised to either radiation treatment arm (LDR brachytherapy or SBRT) an onward referral should be made to the trial team at the Royal Surrey County Hospital. Written patient information on the trial can be provided to the patient before meeting the trial team. Should the patient have a preference for which treatment arm they favour, then they will be offered this as standard of care (if they be deemed suitable by the treating clinician). If patients are willing to have either LDR brachytherapy or SBRT treatment, then they will undergo screening at their first trial appointment.

All men within the trial will have a histological diagnosis of low to intermediate risk prostate cancer defined using National Institute for Health and Care Excellence (NICE) criteria. Those that meet the inclusion criteria as documented in the protocol summary will undergo a baseline urinary flow rate assessment, transrectal ultrasound, and International Prostate Symptom Score (IPSS) questionnaire to ensure they are candidates for the study. All of these screening tests will take place during their first trial appointment at the Stokes Centre for Urology at the Royal Surrey County Hospital. The urinary flow rate should be above 10ml / second, as a figure less than this is suggestive of an obstructive prostate, likely requiring intervention such as a transurethral resection of the prostate (TURP).

A transrectal ultrasound is an important diagnostic tool as it demonstrates the size and shape of the prostate. Men with a prostate gland larger than 60 cc, or those with a large median lobe are not good candidates for LDR brachytherapy and therefore are excluded from the trial, due to challenging dose distribution and increased risk of toxicity.

A Prostate Specific Antigen (PSA) within 60 days of randomisation is required to be used as a baseline result. Any patients deemed high risk and therefore requiring hormonal treatment, as per local policy, alongside their radiotherapy, will be excluded from the study. Patients not eligible for the trial, will be offered an alternative standard of care option and these patients will not be included in the final analysis.

Baseline data include all variables related to demography, assessment for radiotherapy (RT), and eligibility criteria and/or outcomes analyses. In total 134 baseline variables will be collected.

Baseline patient characteristics are assessed during the local Multi Disciplinary Team (MDT) and participant information recorded in 6 data collection instruments (DCI). The baseline DCI capture demography, prior urological procedures, past medical history, urodynamics results and Patient Reported Outcomes Measures (PROMS) collected by means of the Expanded Prostate Index Composite (EPIC-26), the IPSS, International Index of Erectile Function (IIEF-5), and Vaizey Faecal Incontinence score. Treatment allocation takes place once eligibility criteria entered in the baseline DCI are met. The treatment date and treatment visit-related information is gathered followed by an initial assessment at 4 weeks after treatment for PROMs, treatment-related complications, concomitant medications or treatments and of urinary catheter use. Thereafter follow-up assessments include PROMs, blood PSA measurements, clinical or radiographic evidence of tumour progression, use of salvage therapy, and treatment-related complications or any additional medical or surgical treatment. Individual DCIs are used for detail of complications, use of concomitant medications or surgical treatment, withdrawal, and for follow-up after further cancer therapy.

SBRT Radiotherapy planning The prescription dose is 36.25 Gy given in 5 fractions over 1-2 weeks (i.e. daily or alternate daily at department discretion) delivered on linear accelerator. All patients will be recommended to have fiducial markers inserted prior to their treatment. Gold Anchor fiducial markers (Naslund Medical) will be inserted at the same appointment as the Barrigel rectal spacer insertion, to limit appointment burden and anaesthetic for each patient. An added advantage of using Gold anchor markers is their unique design allows a thin needle (22-25G) for implantation, minimising trauma and therefore allowing the patient's planning computerised tomography (CT) scan to be expedited. This will therefore speed up the treatment pathway and reduce appointment burden.

The clinical target volume (CTV) for low-risk patients (Gleason score ≤ 6, T1-T2a or PSA <10 ng/ml) is the prostate only. For intermediate-risk patients (Gleason score 3 + 4, T2b or T2c or PSA 10-20 ng/ml) the CTV is the prostate plus a proximal 1 cm of seminal vesicles from insertion point in the superior-inferior plane. The Planning Target Volume (PTV) is defined as the CTV plus a 5 mm isotropic margin with the exception of a 3mm post margin.

4D Brachytherapy

An outpatient assessment scan conducted prior to procedure determines the size of the prostate and shape using Trans Rectal Ultra Sound (TRUS) in the left lateral position. Five measurements are taken (prostate height, width, length and two para-sagittal lengths). Using the five prostatic measurements, a web-based nomogram calculates how many stranded and loose seeds will be required, which can then be ordered online. The stranded seeds are delivered in preloaded needles numbered in the correct order for implantation. The loose seeds are preloaded into Mick cartridges. Seed implantation performed under general or spinal anaesthesia will follow the protocol guidelines. All patients will undergo a post-implant CT scan for quality assurance within 24 hours to obtain early dosimetric feedback. Post-operative dosimetry aims for the prescription dose of 145Gy are:

* V100% > 90%
* V150% = 35 to 65%
* D90% > 100%
* Urethra V150% < 10%
* Urethra D10% < 150%
* Urethra D30% < 130%
* Urethra Mean < 125%
* Rectum D2cc < 100%
* Rectum D0.1cc < 200Gy

Hyaluronic Acid - Barrigel - rectal spacer Rectal spacing gels have been studied for several years in their addition to radiation treatment for prostate cancer to help reduce radiotherapy toxicities . They act as a barrier between the prostate and the patient's anterior rectum, to absorb unwanted exit dose from the prostate radiotherapy. Barrigel, is a bio-degradable natural gel product. The spacer gel is inserted between the anterior rectal wall and the prostate, known as Denonvilliers' fascia, to temporarily position the anterior rectal wall away from the prostate during radiotherapy for prostate cancer. The gel is slowly absorbed over 1-3 years, ensuring the prostate remains in a similar position for the treatment delivery. To ameliorate the radiation effect on rectal tissue, all SBRT and LDR Brachytherapy patients will undergo transperineal application of a Barrigel rectal spacer. Barrigel will be inserted under ultrasound guidance, by trained professionals using an aseptic technique. The gel can be inserted under local or general anaesthetic. For patients receiving SBRT treatment, no general anaesthesia is required in their treatment work up and therefore Barrigel will be inserted into Denonvilliers' fascia under local anaesthetic following fiducial marker insertion. For patients receiving LDR brachytherapy, the gel will be inserted once all the radioactive seeds have been inserted during the same procedure. All patients will have at least 3ml of Barrigel inserted into Denonvilliers' space, aiming to create 1cm separation from the prostate base to its apex from the anterior rectal wall. For intermediate risk SBRT patients, who will have the first 1cm of seminal vesicle included within the CTV, additional Barrigel to create 1cm separation from the seminal vesicle to the anterior rectal wall will be added. The gel will be inserted centrally, aiming for a symmetrical distribution on each side of the prostate under trans-rectal ultrasound supervision. Both sagittal and axial views on ultrasound should be assessed to check midline symmetry and adequate placement from base to apex, aiming for at least 1cm separation.

It is well documented that radiation toxicities are typically at their worst within the first 3 months following treatment. Patients will therefore have an intensive follow up period following their respective treatments to assess toxicity. Their end of treatment date will be noted as their Day 0 with their first follow up appointment 4 weeks later. Within the first 3 months following treatment they will have 2 telephone consultations (at week 4 and week 8) in which they will have Common Terminology Criteria for Adverse Events (CTCAE) scoring assessment of their side effects and will complete the PROMS questionnaires. The patient will then have a face-to-face appointment at 3 months. If the patient underwent SBRT treatment their follow up will be with the treating Oncologist. If the patient underwent brachytherapy they will be followed up by the brachytherapy team at the Stokes Centre. The patients first PSA will be recorded at 3 months after Day 0. The interval between follow up appointments will increase after the 3-month period as the acute toxicities wear off however unscheduled appointments can be booked if required.

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥18 years at randomisation
* The research subject must have capacity to sign a written informed consent document for the trial
* WHO performance status 0 - 2
* Gleason score 3+3 or 3+4
* PSA ≤ 20 ng/ml (please note if the treating clinician determines androgen deprivation therapy (ADT) is required this is an exclusion criteria). A PSA must be available within 60 days of randomisation.
* Clinical and/or MRI stage T1c -T2c, N0-X, M0-X
* Histological confirmation of prostate adenocarcinoma within the last 18 months (unless on active surveillance). Patients who were on active surveillance should have an up-to-date MRI within 8 weeks of the decision to treat to confirm organ confined disease.

Exclusion Criteria:

* Previous malignancy within the last 2 years (except basal cell carcinoma or squamous cell carcinoma of the skin), or if previous malignancy is expected to significantly compromise 10-year survival.
* Patients under investigation for synchronous primary at time of randomisation
* Prior pelvic radiotherapy.
* Prior treatment with ADT or current need for ADT based on risk features

  * Prostate cancer in greater than 50% of template biopsy cores or a significant maximum core length containing prostate cancer for which the treating clinician deems the patient would benefit from ADT
* Any prior active treatment for prostate cancer (patients previously on active surveillance are eligible if they meet all other eligibility criteria)
* Life expectancy < 10 years Men with a prostate gland larger than 60 cc, or those with a large median lobe• Hip prostheses or any other implants/hardware that introduce substantial CT artefacts making it challenging to delineate the target or organs at risk. This is to be assessed on a case-by-case basis with the available staging imaging.
* Medical conditions likely to make radiotherapy inadvisable e.g. inflammatory bowel disease, significant urinary symptoms.
* International Prostate Symptom Score (IPSS) > 15 points
* Anticoagulation with warfarin/ bleeding tendency making fiducial placement, spacer gel insertion or brachytherapy unsafe in the opinion of the clinician
* Contraindications for Barrigel insertion such as previous documented allergic reaction to gel, previous rectal surgery or known rectal fistula.
* Participation in another concurrent treatment protocol for prostate cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
EPIC-26 score minimally important difference | Scores will be collected pre-treatment, 1, 2, 3, 6, 12, 18, and 24 months after treatment, and then yearly up to the 5-year post-treatment time point.
  The EPIC-26 questionnaire is a preeminent tool extensively characterised to measure health-related quality of life in men with localised prostate cancer. Our study is powered to detect the minimally important differences in urinary, sexual, and bowel function domains relative to the pre-treatment values.

SECONDARY OUTCOMES:
International Prostate Symptom Score (IPSS) | Scores will be collected pre-treatment and at 1, 2, 3, 6, 12, 18, and 24 months after treatment, and then annually up to the 5-year post treatment time point.
  IPSS assesses urinary voiding symptoms and bother. For voiding symptoms, a score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms, and the urinary bother scale ranges from 0 (Delighted) to 6 (Terrible).
International Index of Erectile Function (IIEF-5) | Scores will be collected pre-treatment and at 1, 2, 3, 6, 12, 18, and 24 months after treatment, and then annually up to the 5-year post treatment time point.
  The IIEF-5, also known as the Sexual Health Inventory for Men (SHIM) score , characterises the severity of erectile dysfunction (ED) with lower scores indicating greater dysfunction (5-7 severe, 8-11 moderate, 12-16 mild-to-moderate, 17-21 mild, 22-25 no ED).
Vaizey faecal inconticence score | Scores will be collected pre-treatment and at 1, 2, 3, 6, 12, 18, and 24 months after treatment, and then annually up to the 5-year post treatment time point.
  The Vaizey Incontinence Score is a general-purpose scale for faecal incontinence that ranges from 0 to 24 with higher scores representing worst incontinence.

OTHER OUTCOMES:
Prostate-Specific Antigen (PSA) | Values will be collected pre-treatment, at 3 and 6 months post-treatment, and thereafter every 6 months up to the 5 years time point.
  PSA - 3 consecutive PSA rises within the first 2 years post treatment or a PSA rise of 2 ng/mL or more from the patient's nadir result after the 4 year time point will be deemed as biochemical failure and warrants further re-staging investigations. Patients will be kept on follow up for the 5 year follow up period, if appropriate, despite biochemical failure, to account for late PSA bounces .
Survival | 5 years post-treatment.
  Survival outcomes are time-to-event variables i.e. relapse-free survival, cancer-specific survival, and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Langley, Professor of Urology, Study Chair — Royal Surrey NHS Foundation Trust
Locations (1):
- Royal Surrey NHS Foundation Trust, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Unsure how rules apply to non US trials.Need more specific information.

REFERENCES:
- [Background] Vaizey CJ, Carapeti E, Cahill JA, Kamm MA. Prospective comparison of faecal incontinence grading systems. Gut. 1999 Jan;44(1):77-80. doi: 10.1136/gut.44.1.77. PMID 9862829
- [Background] Mariados NF, Orio PF 3rd, Schiffman Z, Van TJ, Engelman A, Nurani R, Kurtzman SM, Lopez E, Chao M, Boike TP, Martinez AA, Gejerman G, Lederer J, Sylvester JE, Bell G, Rivera D, Shore N, Miller K, Sinayuk B, Steinberg ML, Low DA, Kishan AU, King MT. Hyaluronic Acid Spacer for Hypofractionated Prostate Radiation Therapy: A Randomized Clinical Trial. JAMA Oncol. 2023 Apr 1;9(4):511-518. doi: 10.1001/jamaoncol.2022.7592. PMID 36757690
- [Background] Langley SE, Laing RW. 4D Brachytherapy, a novel real-time prostate brachytherapy technique using stranded and loose seeds. BJU Int. 2012 Feb;109 Suppl 1:1-6. doi: 10.1111/j.1464-410X.2011.10824.x. PMID 22239223
- [Background] Alexander SE, Kinsella J, McNair HA, Tree AC. National survey of fiducial marker insertion for prostate image guided radiotherapy. Radiography (Lond). 2018 Nov;24(4):275-282. doi: 10.1016/j.radi.2018.06.003. Epub 2018 Jul 7. PMID 30292494
- [Background] Tree AC, Ostler P, van der Voet H, Chu W, Loblaw A, Ford D, Tolan S, Jain S, Martin A, Staffurth J, Armstrong J, Camilleri P, Kancherla K, Frew J, Chan A, Dayes IS, Duffton A, Brand DH, Henderson D, Morrison K, Brown S, Pugh J, Burnett S, Mahmud M, Hinder V, Naismith O, Hall E, van As N; PACE Trial Investigators. Intensity-modulated radiotherapy versus stereotactic body radiotherapy for prostate cancer (PACE-B): 2-year toxicity results from an open-label, randomised, phase 3, non-inferiority trial. Lancet Oncol. 2022 Oct;23(10):1308-1320. doi: 10.1016/S1470-2045(22)00517-4. Epub 2022 Sep 13. PMID 36113498
- [Background] van As N, Yasar B, Griffin C, Patel J, Tree AC, Ostler P, van der Voet H, Ford D, Tolan S, Wells P, Mahmood R, Winkler M, Chan A, Thompson A, Ogden C, Naismith O, Pugh J, Manning G, Brown S, Burnett S, Hall E. Radical Prostatectomy Versus Stereotactic Radiotherapy for Clinically Localised Prostate Cancer: Results of the PACE-A Randomised Trial. Eur Urol. 2024 Dec;86(6):566-576. doi: 10.1016/j.eururo.2024.08.030. Epub 2024 Sep 11. PMID 39266383
- See also: NICE Prostate cancer: diagnosis and treatment — https://www.nice.org.uk/guidance/ng131
- See also: 4D Brachytherapy practical guide — https://bxta.com/uk/healthcare-professionals/4d-brachytherapy/a-practical-guide-to-4d-brachytherapy/
- See also: IPSS questionnaire — https://prostate.ie/wp-content/uploads/IPSS.pdf
- See also: IIEF-5/SHIM questionnaire — https://www.baus.org.uk/_userfiles/pages/files/patients/leaflets/SHIM.pdf